CLINICAL TRIAL: NCT06795620
Title: Tolerance Study of Allogeneic of Adipose Tissue Derived Mesenchymal Stroma/Stem Cells (AdMSC) Transplantation in Patients With Critical Limb Ischemia.
Acronym: AlloDREAM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0168; 2023-509312-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-16; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Critical Limb Ischemia
Keywords: Adipose tissue; allogeneic AdMSC; cell therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CellReady (Experimental): All the patients will be included and will have AdMSC injections (CellReady®) in their ischemic led. They will be follow-up during 6 months.
  Interventions: Drug: Adipose tissue derived mesenchymal Stroma/stem Cells transplantation

INTERVENTIONS:
Drug: Adipose tissue derived mesenchymal Stroma/stem Cells transplantation — Allogeneic adipose tissue-derived stromal cells (AdMSC) (CellReady ® drug) will be administered intramuscularly into the ischemic limb (dose of 90x10^6 AdMSC) of patients. They will be followed at 1 day, 7 days, 30 days, 90 days, and 180 days after the injection.

SUMMARY:
Critical limb ischemia (CLI) is the most severe stage of peripheral arterial disease (PAD). Cell therapy delivered to the ischemic muscle constitutes a promising approach to treat CLI patients with no or poor options of vascularization. Pre-clinical study and clinical phase I have demonstrated the safety and feasibility of the use of autologous AdMSC treatment in patients without option for revascularization CLI patients and encouraging preliminary efficacy results have been highlighted in the pilot phase. In order to optimize AdMSC quality and to accelerate treatment availability researchers decide to test the use of allogeneic cryopreserved AdMSC from healthy donor. The aim of this phase I study is to evaluate the safety of allogeneic AdMSC injection in ischemic leg.

DETAILED DESCRIPTION:
Lower limbs arteries are a frequent localization of atheroma in elderly people (15-20% after 70 years). The most severe stage of the disease, critical limb ischemia (CLI), defined clinically by the presence of rest pain or ischemic ulcer with an ankle pressure <50 mmHg or a toe pressure <30 mmHg or a TcPO2 <30 mmHg, has a dramatic prognosis at 12 months, with 30% of the patients alive with an amputation, 20% mortality and only 20% of patients with a resolved disease, independently from the treatment. The only validated treatment for this disease is revascularization by endovascular procedures or open surgery. Patients with no option or poor option (high risk) for revascularization have the worst prognosis. Regenerative medicine has been studied in this field, by the injection of bone marrow derived stem cells in the ischemic limb to improve neo-angiogenesis. Despite the encouraging first results, few studies have shown a clinical interest of this kind of approach. The products tested were heterogeneous compounds derived from the bone marrow.

Different types of stem cells have recently been studied in clinical trial on ischemic disease of the heart and muscular arteries. Adipose derived stem cell, have shown in vitro and in vivo models a stronger potential of success in recovering from ischemic disease and oxygenation of the tissues.

Scientists already shown in a phase I study, that adipose derived mesenchymal cells injected in patients with CLI and no option for revascularization, had a very good tolerance and interesting effects on skin oxygenation and healing.

In order to optimize the quality of the AdMSC, to avoid the abdominal sample under anesthesia in the already suffering patients and to have the cellular product available quickly, without waiting the 15 days of culture, researchers envisage the use of AdMSC of allogeneic origin taken from healthy donors and cryopreserved after culture. Indeed, the results of phase 1 of ACellDREAM showed that almost half of the patients suffering from IC had to be amputated during the 15 days of culture. Preliminary experiments show that the phenotypic characteristics, in vitro properties and in vivo biodistribution of these cells after freezing are unchanged.

Researchers are planning a single phase, phase I study to evaluate the tolerability of intramuscular injection of allogeneic AUC in patients with critical non-revascularizable ischemia, or with persistent ischemia despite revascularization.

The aim of this phase I is to evaluate safety of allogeneic AdMSC transplantation in patients with critical limb ischemia with poor options or no option for revascularization. Ten patients will be included and have AdMSC injection in their ischemic leg. Patients will be follow-up during six months to evaluate ulcer evolution, wound healing, pain, blood flow and immune response in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old,
* Patients with CLI according international definition: 1) rest pain of ischemic origin or ischemic trophic disorder present for at least 15 days, and 2) an ankle pressure ≤50 mmHg (≤70 mmHg for diabetic patients) or a toe pressure ≤30 mmHg or a TcPO2 ≤30 mmHg,
* Patient not revascularizable by decision of the surgeon or anesthesiologist orpatient with persistent critical ischemia after revascularization,
* Patient with a life expectancy greater than 6 months,
* Patients who signed the informed consent,
* Women of childbearing age with effective contraception (oral contraception, IUD, dermal implant) and with negative pregnancy test,
* Patient affiliated to a social security system.

Exclusion Criteria:

* Need of a major amputation (amputation at or above the ankle) within 1 month following the inclusion,
* Another clinical trial participation (except observational studies),
* Patient with active cancer history in the 5 previous years except cured basal cell carcinoma or cured low-stage melanoma,
* Patient allergic to local anesthetics
* Immunosuppressive therapy
* Ulcers with exposure of tendons, osteomyelitis, or clinically uncontrolled infection,
* Patient under the protection of justice or under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the tolerance | 6 months
  local and systemic tolerance during 6 months by the collection and analysis of adverse events (serious or non-serious) throughout the duration of the study

SECONDARY OUTCOMES:
Evaluation of the efficacy of the treatment on critical limb ischemia. | Day 30, Day 90, and Day 180
  Proportion of patients without criteria of CLI
Evaluation of the evolution of ischemia objective parameters. | Day 0, Day 30, Day 90, and Day 180
  Pressures, laser-Doppler and TcPO2
Evaluation of the healing. | Day 30, Day 90, and Day 180
  Number of complete scarring
Evaluation of the proportion of patients who required a major amputation. | Day 180
Evaluation of the pain Evolution | Day 0, Day 7, Day 30, Day 90, and Day 180
  VAS (visual analogue scale), consumption of morphine or non-morphine analgesics
Evaluation of the neovascularization on the treated leg. | Day 30, Day 90, and Day 180
  Determination of the number of neo-vessels formed by angiography, angio Magnetic resonance imaging (MRI) or angio-scanner.
Evaluation of the proportion of patients included who had all the injections. | Day 0
Evaluation of the evolution of the quality of life | Day 0, Day 30, Day 90, and Day 180
  Claudication Scale (CLAU-S®)
Evaluation of the security. | Day 0, Day 1, Day 7, Day 30, Day 90, and Day 180
  Description of all adverse reaction during the trial
Evaluation of the immunomodulatory activity of the injected cells. | Evaluated at Day 1, Day 7, Day 30, Day 90, and Day 180
  - Immuno-monitoring by evaluation of the different circulating immune populations (Th1, Th2, Th17, Treg ...) associated with functional tests in vitro and immunological assays of pro and anti-inflammatory cytokines (IL-1, IL-2, IL-4, IL-6, IL-10, IL-12, TNFα, IFNγ).
Evaluation of the patient's immune response against Adipose-derived mesenchymal stem cells (AdMSCs) | Day 30
  Dosage of anti HLA (human leukocyte antigen) donor antobodies.
Evaluation of the evolution of the quality of life. | Day 0, Day 30, Day 90, and Day 180
  EuroQol (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier LAPEBIE, Dr, Principal Investigator — Service de Médecine Vasculaire, Hôpital Rangueil, CHU de Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No